CLINICAL TRIAL: NCT03320668
Title: Efficacy of the Otago Exercise Program (OEP) Delivered as Group Training Versus Individually Tailored Training in Community-dwelling Adults Between 65 and 80 Years Old
Brief Title: Efficacy of the Otago Exercise Program Delivered as Group Training Versus Individually Tailored Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Salud Carlos III (Other Government)
Collaborators: Fondo de Investigacion Sanitaria (Other); Osakidetza (Other); MurciaSalud (Other Government)
Responsible Party: Principal Investigator, Teresa Moreno Casbas, Unit Director, Instituto de Salud Carlos III
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI16CIII/00031
Record Dates: First submitted 2017-10-20; First posted 2017-10-25 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Age Problem
Keywords: Falls Prevention; Otago Program; Community-Dwelling

STUDY DESIGN:
Intervention Model Description: Non-inferiority clinical trial, multicentric, simple blind
Who Masked: Outcomes Assessor
Masking Description: Blind analysis to prevent bias
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual OEP (No Intervention): Randomized subjects (65 to 80-year-old) receiving individual Otago Exercise Program (OEP) training in a total of nine Primary Care Centers.
  An "OEP leader" trained nurse/physiotherapist will perform in its community consult individual education to each participant in five sessions: In the 1st, 2nd, 4th and 8th week and one reinforcement session after six months. A telephone call to each participant (following a predefined telephonic interview protocol) will be carried out in the months without training session to perform the follow-up.
- Group OEP (Experimental): 65-80 year-old randomized subjects receiving group Otago Exercise Program (OEP) training in a total of nine Primary Care Centers.
  Interventions: Other: Otago Exercise Program (OEP)

INTERVENTIONS:
Other: Otago Exercise Program (OEP) — A nurse/physiotherapist supported by an "instructor"-trained professional will give Otago Exercise Program (OEP) education to 10-people groups in 5 sessions (1st, 2nd, 4th and 8th week and one reinforcement session after 6 months). Telephone calls to participants will be made during non-training months (following a predefined telephonic interview protocol) to follow up. The OEP reduces the number of falls and fall-related injuries, improving balance and strength, confidence in performing everyday activities without falling. Whilst it has been shown to be effective in 4 controlled trials in New Zealand, it has not been tested in a primary care setting in Spain for feasibility, impact, acceptability and cost-effectiveness.
  Other Names: Usual Practice
  Arms: Group OEP

SUMMARY:
A non-inferiority controlled clinical trial using randomization for allocation at the level of general practice in 21 centers (in 8 Spanish regions), to compare a group Otago exercise program (OEP) [delivered by specifically trained instructors and supplemented by prescriptive recommendations for home exercising], with an individual OEP [also delivered by specifically trained professionals and supplemented by prescriptive recommendations for home exercising], with twelve months follow-up to determine the effectiveness of the OEP in terms of prevention of falls in a community-dwelling 65- to 80-year-old population.

DETAILED DESCRIPTION:
OBJECTIVES:

To compare the effectiveness of the Otago Exercise Program (OEP) delivered as group training versus individually tailored training in community-dwelling adults between 65 and 80 years old, on the probability of falls, improved functional balance and muscle strength and, quality of walk in the 12 months follow up.

To compare the effectiveness of both interventions to improve dynamic and static balance and gait quality in the same population.

DESIGN:

Non-inferiority clinical trial, multicentric, simple blind (blind analysis to prevent bias), with two interventions, implementation of group and individual OEP with random assign. The follow-up period will be twelve months after the OEP training.

FIELD OF STUDY:

21 Primary Health Centers (PHC) belonging to the National Health System in 8 different regions: Andalucía, Asturias, Islas Baleares, Canarias, Cataluña, Comunidad de Madrid, Región de Murcia and País Vasco

PARTICIPANTS:

Subjects who belong to primary care centers in the same health area, 65 to 80 years of age, who are not institutionalized, independent for walk (the score of the first part of the Short Physical Performance Battery scale (SPPB scale) in relation to balancing must be different from zero in any assessed position) and provide informed consent to participate in the study.

VARIABLES OF STUDY:

Principal Outcome: Percentage of falls (percentage of subjects falling)

Other Outcomes:

Safety of Intervention; Feasibility of interventions; Feasibility of the cascade training model based on the OEP; Economic analysis and added therapeutic value of both interventions.

DATA COLLECTION:

Subjects will be selected from the health centers through active recruitment by the health professionals.

The recruitment will be consecutive among the patients in the agenda in the days between 10 to 19 of each month from September 2017-December 2018.

Data will be collected at month 0, 6 and 12. Randomization will be performed by PHC and by subjects.

DATA ANALYSIS:

A descriptive analysis of sociodemographic and fall variables will be performed. The analysis to the comparative data between the two groups of the Randomize Clinical Trial will be done by protocol. In addition, an analysis will be made for the incidence density of falls, using Poisson regression models. For all a confidence level of 95% will be assumed, and the statistical software to be used to carry out the analysis will be Statistical Package for the Social Sciences version 22 (SPSS v22).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who belong (ascribed) to primary healthcare centers of the same health area, aged 65 to 80 years, non-institutionalized, independents for ambulation (the scores achieved from the first part of SPPB scale in relation of the balance will be different from zero in any position evaluated.) and provide their informed consent for participating in the study.

Exclusion Criteria:

* Subject such residential period in the Health Basic Area of the primary health center or it life expectancies has lower 9 months. in the health area of the primary healthcare center.
* Mild and moderate cognitive impairment (according to the diagnosis from medical history).
* Sight-impairment or hearing impairment which prevent to follow the intervention (according to the diagnosis from medical history).
* Absolute contraindication to perform physical exercise (according to the diagnosis from medical history)

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 878 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Percentage of falls | 12 months
  The participant will be provided with a notebook which should be completed each month. In the case a fall occur, the patient will be asked to fill the following items regarding the fall characteristics: Data, place, context in which the fall happened, consequences and attention required.

SECONDARY OUTCOMES:
Adverse events | 12 months
  1. Adverse events during the intervention related to exclusion criteria (indication for a subject to leave the project)
  2. Adverse effects which can be directly or potentially associated with Otago exercises. For that, it will be established an external committee which will classify the adverse event among related, potentially related and none related with Otago exercise execution.
Adherence | 12 months
  Adherence level to exercise program will be measured following the Exercise Adherence Rating Scale (EARS) through self-declared falls diary.
  The EARS questionnaire is composed of 6 items, each of them is scaled from 0 (minimum) to 4 (maximum score). Total score is the sum of the 6 items, so that it ranges from a minimum score of 0 and a maximum score of 64.
  Adherence measurements will be collected at 6 and 12 months.
Participant satisfaction | 12 months
  Participant satisfaction with the intervention will be measured through "ad hoc" survey which include the following items:
  4.1. Received information about exercise program and its benefits 4.2. Received Training about Otago Exercise Program 4.3. Assessment of Material 4.4. Teaching skills of your OEP trainer 4.5. Receptiveness of your health care professional to solve your doubts about the OEP 4.6. Global satisfaction with Otago Exercise Program
  Each item will be scaled from 0 (Totally unsatisfied) to 4 (Very satisfied).
  Total minimum and maximum scores are 0 and 64, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Moreno-Cascas, Doctor, Study Director — Instituto de Salud Carlos III
Locations (9):
- Spain (9):
  - Osakidetza, Vitoria-Gasteiz, Araba Kalea, 45, Vitoria-Gasteiz
  - Universidad de Córdoba, Córdoba, Av. de Medina Azahara, 5
  - Servicio de Salud de Madrid, Madrid, Avenida Abrantes, 55
  - Servicio de Salud de Canarias, Las Palmas de Gran Canaria, Avenida Juan Xxiii,17
  - Servicio Murciano de Salud, Murcia, Calle Central, 7, Espinardo
  - Servei de Salut de Les Illes Balears, Palma de Mallorca, Carrer de La Reina Esclaramunda, 9, Palma
  - Institut Català de la Salut (ICS), Barcelona, Gran Via de Les Corts Catalanes, 587-589
  - Institut Català de la Salut, Barcelona, Gran Via de Les Corts Catalanes, 587-589
  - Servicio de Salud del Principado de Asturias, Oviedo, Plaza Del Carbayón, Oviedo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Albornos-Munoz L, Blanco-Blanco J, Cidoncha-Moreno MA, Abad-Corpa E, Rivera-Alvarez A, Lopez-Pisa RM, Caperos JM; Otago Project Working Group Consortium; Moreno-Casbas MT. Efficacy of the Otago-Exercise-Programme to reduce falls in community-dwelling adults aged 65-80 when delivered as group or individual training: Non-inferiority-clinical-trial. BMC Nurs. 2024 Oct 1;23(1):705. doi: 10.1186/s12912-024-02310-3. PMID 39354514
- [Derived] Angeles CM, Laura AM, Consuelo CM, Manuel RR, Eva AC, Covadonga GA; Otago Project Working Group. The effect that the Otago Exercise Programme had on fear of falling in community dwellers aged 65-80 and associated factors. Arch Gerontol Geriatr. 2022 Mar-Apr;99:104620. doi: 10.1016/j.archger.2022.104620. Epub 2022 Jan 4. PMID 34999543